CLINICAL TRIAL: NCT04637724
Title: Transcranial Weak Current Stimulation Treatments for Working Memory Dysfunction in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oded Meiron (Other)
Responsible Party: Sponsor-Investigator, Oded Meiron, Director of Non-invasive Brain Stimulation Clinic, Herzog Hospital
Organization: Herzog Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 337-19
Record Dates: First submitted 2020-11-11; First posted 2020-11-20 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia; Schizo Affective Disorder
Keywords: Working memory; Schizophrenia symtom severity,; Prefrontal tDCS; Event related EEG
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Active tDCS versus Sham tDCS intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Experimental): active prefrotal tDCS: 20 mins pes tDCS session, twice a day for 5 days. Total of 10 ative tDCS sessions.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): Sham prefrontal tDCS: sham stimulation 20 mins per session, twice a day for 5 days. Total of 10 sham stimulation sessions
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — 10 sessions of Anodal tDCS of the dorsolateral prefrontal cortex over a period of 5 consecutive days (two session a day). Each session includes the placement of two tDCS electrodes (anodal at left prefrontal area and cathodal above the vertex) and 20 mins of anodal prefrontal stimulation. The tDCS session is received two time a day with a 3-5 hours interveal betwen sessions.
  Other Names: Prefrontal tDCS

SUMMARY:
For the present study, Investigators will examine the efficacy of active prefrontal anodal tDCS versus placebo (sham) interventions to treat WM dysfunction in schizophrenia.

Investigators selected the prefrontal stimulation modality that proved most effective in enhancing high-load WM performance in single dose stimulation in healthy participants . The study employs a multi-stimulation approach, with 2 sessions per day for 5 consecutive days in the active treatment group (n=15) compared to a group that receives only sham stimulation (n=15). This preliminary approach is based upon findings of a recent study applying cathodal tDCS stimulation over left temporoparietal cortex (with left prefrontal anodal stimulation) for the treatment of persistent auditory hallucinations in schizophrenia. In a a recent study clinical benefits were maintained for at least 3 months following stimulation. In the present study, in addition to clinical outcome, researchers will evaluate whether similar improvement can be obtained with WM, EEG activity, and functional outcome (e.g., discharged from hospitalization following significant improvement or remission).

DETAILED DESCRIPTION:
In a recent tDCS study investigators conducted with 41 healthy participants, researchers administered a single blind tDCS protocol that included an active unilateral DLPFC condition (2 mA for 15 minutes, anode over the left DLPFC (midpoint between F3-AF3) and cathode over the dorsal area of the superior parietal cortex (at Cz) versus a sham condition to investigate changes in online working memory function. Our preliminary tDCS results indicated gender-dependent (left enhancement in males versus females) high-load WM enhancement during active prefrontal stimulation versus sham stimulation. The observed prefrontal tDCS enhancing effect on high-load WM function indicated that left DLPFC tDCS could be implemented with SZP who suffer from inefficient left DLPFC engagement during medium to high-load WM maintenance.

Given the lack of effective treatments for attenuating WM impairments and the importance of these impairments to functional outcome in schizophrenia, tDCS based cognitive-enhancing approaches may become an important new treatment method, which will consequently improve treatment and functional outcome in schizophrenia patients.The innovative nature of the study's proposed research project is that it promotes non-invasive focal (left prefrontal cortex) neuromodulation to improve cognitive functioning as well as illness severity in SZP. Most importantly, unlike antipsychotic medication that affects the entire brain circuitry and produces undesired side effects (e.g., extrapyramidal effects, weight gain, hyperlipidemia, and sexual dysfunction), the current non-invasive focal intervention is aimed at reducing specific prefrontal dysfunctions in schizophrenia by specific targeting of prefrontal electrophysiological disturbances (e.g., frontal theta synchrony) within regions known to regulate behavior and the consolidation of goal-directed information.

Hypothesis Essentially, currently proposed tDCS treatment is hypothesized to improve working memory functioning and reduce symptom severity in people diagnosed with schizophrenia versus sham prefrontal tDCS (placebo).The theoretical premise for our prediction implies that effective inhibition of excessive dopaminergic mesolimbic activity (impaired in schizophrenia), could result from excitatory left-prefrontal tDCS, which has been shown to increase executive regulation of behavior in healthy individuals and people diagnosed with schizophrenia .

Research plan outline For the present study, investigators will examine the efficacy of active prefrontal anodal tDCS versus placebo (sham) interventions to treat WM dysfunction in schizophrenia. Investigatros selected the prefrontal stimulation modality that proved most effective in enhancing high-load WM performance in single dose stimulation in healthy participants. A multi-stimulation approach is implemnted, with 2 sessions per day for 5 consecutive days in the active treatment group (n=15) compared to a group that receives only sham stimulation (n=15). This preliminary approach is based upon findings of a recent study applying cathodal tDCS stimulation over left temporoparietal cortex (with left prefrontal anodal stimulation) for the treatment of persistent auditory hallucinations in schizophrenia . In a recent study clinical benefits were maintained for at least 3 months following stimulation. In the present study, in addition to clinical outcome, we will evaluate whether similar improvement can be obtained with WM, EEG activity, and functional outcome (e.g., discharged from hospitalization following significant improvement or remission).

In regards to efficacy, since WM is considered a core cognitive deficit in schizophrenia, investigators will monitor working memory, psychosis severity and global outcome, at baseline, immediately following tDCS intervention, and at 1, 4, and 8, 12, and 16 week intervals, following the termination the five-day treatment. Importantly, in order to show external validity of our efficacy analysis we will examine functional outcome (level of independence), six months after the termination of the tDCS intervention.

Finally, since DLPFC stimulation may contribute to long-term electroencephalography (EEG) theta- rhythm functional connectivity, associated with increased large-scale theta synchronization, WM function, and episodic memory formation, investigatros will examine effects of tDCS on prefrontal versus whole-brain EEG theta activity obtained during a WM task (see verbal n-Back task), using event-related potential (ERP) and event-related spectral power (ERSP) techniques similar to those in used in recent EEG studies in schizphrenia patients. Demonstrating significant functional-connectivity EEG differences in responders versus non-responders from baseline to post-intervention measurements will significantly increase the validity of our proposed prefrontal pathophysiological mechanism as significantly impacting psychosis severity and clinical outcome in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75
* Primary diagnosis of DSM-IV schizophrenia (including schizoaffective disorder)
* Right handed
* Under stable doses of antipsychotic medication for ≥4 weeks
* Normal vision by self report and physical exam
* Use of effective method of birth control for women of childbearing capacity
* Willing/capacity to provide informed consent
* Outpatients or volunteering inpatients or involuntary patients with consent of legal guardian.

Exclusion Criteria:

* Current or past history of substance dependence or abuse (excluding nicotine)
* Other current Axis I disorders
* History of seizure, epilepsy in self or first degree relatives, stoke, brain surgery, head injury, intracranial metal implants, known structural brain lesion, devices that may be affected by tDCS (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Frequent and persistent migraines
* History of adverse reaction to neurostimulation
* Participation in study of investigational medication within 6 weeks
* Pregnancy
* Women who are breast-feeding
* Current significant laboratory abnormality

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
change in Positivie and Negative Syndrome Scale (PANSS, minimum score = 30, maximum score = 350, higher score indicate incresed ilness severity, lower scores indicate lower ilness severity) scores from baseline to post-tDCS intervention | Immediately after 10-day tDCS-intervention
  change in total scores of the Positive and negative syndrome scale for Scizophrenia
change in working memory accuracy scores from baseline to post-tDCS intervention | Immediately after 10-day tDCS intervention
  change in verbal working memory accuracy (scores range from 0 to 126 correct responses)
change in working memory reaction times from baseline to post-tDCS intervention | Immediately after 10-day tDCS intervention
  change in mean reaction times of correct rsponses (i.e., hits) (measures in millisecods range from 400 to 2000 msec)

SECONDARY OUTCOMES:
change in Mismatch neagtivity (MMN) event related potentials from baseline to post-tDCS intervention | Imediatly after after 10-dat tDCS intervention
  change in MMN amplitudes from baseline to post-tDCS intervention (change in microVolts: change of 1 to 5 microvolts undet Fz electrode
change from baseline to post-tDCS intervention in Induced EEG theta power folowing verbal command | Immediatly after tDCS intervention
  change in mean theta power activity (e.g., under Fz electrode, absolute power scale: µV2), change in mean absolute power of theta oscillations
change from baseline to post-tDCS intervention in Induced EEG alpha power folowing verbal command | Immediatly after tDCS intervention
  change in mean alpha power activity (e.g., under Fz electrode, absolute power scale: µV2), change in mean absolute power of alpha oscillations

CONTACTS AND LOCATIONS:
Overall Officials: Alex Borochov, MD, Principal Investigator — Herzog Medical Center
Locations (1):
- Herzog Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
non personal coded data indicating the participants change in working memory scores, change in psychosis severiry PANSS scores, and change in MMN amplitudes: comparing active tDCS group versus shham-tDCS group

REFERENCES:
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236
- [Derived] Meiron O, Yaniv A, Rozenberg S, David J. Transcranial direct-current stimulation of the prefrontal cortex enhances working memory and suppresses pathological gamma power elevation in schizophrenia. Expert Rev Neurother. 2024 Feb;24(2):217-226. doi: 10.1080/14737175.2023.2294150. Epub 2024 Feb 6. PMID 38084398
- [Derived] Meiron O, David J, Yaniv A. Left prefrontal transcranial direct-current stimulation reduces symptom-severity and acutely enhances working memory in schizophrenia. Neurosci Lett. 2021 Jun 11;755:135912. doi: 10.1016/j.neulet.2021.135912. Epub 2021 Apr 21. PMID 33894334